CLINICAL TRIAL: NCT03755986
Title: Performance and Usability Evaluation of the Atomo HIV Self-Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Holdsworth House Medical Practice (Other)
Collaborators: Atomo Diagnostics (Unknown)
Responsible Party: Principal Investigator, Dr. Mark Bloch, A/Prof, Holdsworth House Medical Practice
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ARST001-2016
Record Dates: First submitted 2017-02-22; First posted 2018-11-28 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ATOMO Diagnostic Test (Other): All patients will receive an ATOMO diagnostic test to use. There is no comparative arm.
  Interventions: Device: ATOMO Diagnostic Test

INTERVENTIONS:
Device: ATOMO Diagnostic Test — The ATOMO diagnostic test device is the only intervention used in this study.

SUMMARY:
The study seeks to enroll 501+ patients to use a HIV self testing device to test for HIV in a blood sample drawn by finger prick. The purpose of the trial is to assess the usability of the device by providing participants with video and written instructions on how to correctly obtain a result from the device.

ELIGIBILITY:
Inclusion Criteria The inclusion criteria are informed by the indications for HIV testing contained in the National HIV Testing Policy, which states that HIV testing is indicated in the following groups: MSM; people who inject drugs; people with multiple sex partners or recent partner change; people having travelled to countries of high prevalence and engaged in risk behavior; people from high prevalence countries; partners of the above; and partners of people living with HIV infection.

Recruitment will be restricted to people who satisfy the following criteria:

1. Attending health clinic or community-based testing study sites
2. Aged 18 years or more
3. Requesting HIV testing and/or in whom HIV testing is indicated
4. Willing and able to give their own informed consent
5. Willing to participate in and comply with the study procedures

Exclusion Criteria

The following people will be excluded from the study:

1. People in whom HIV testing is not indicated or not appropriate
2. People not fluent in English in whom provision of informed consent or compliance with the study procedures may be problematic
3. People who have participated in the study previously

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Questionnaire scoring each step of performing the self-test | Assessed at one time point per patient (visit 1) approximately 1 hour
  To assess the ability of typical self-test users to follow the test instructions and perform the test accurately and to identify any issues or difficulty they may experience whilst performing the test.
Questionnaire scoring each step of performing the self-test | Assessed at one time point per patient (visit 1) approximately 1 hour
  To assess the ability of typical self-test users to perform the test accurately
Questionnaire scoring each step of performing the self-test | Assessed at one time point per patient (visit 1) approximately 1 hour
  To identify any issues or difficulty the self-test users may experience whilst performing the test.

SECONDARY OUTCOMES:
Questionnaire scoring each step of performing the self-test | Assessed at one time point only per patient (visit 1)approximately 1 hour
  To assess the ability of typical self-test users to follow the test instructions and perform the test accurately when the user knows they did not perform the steps of testing properly in their initial attempt.
Comparison of self-test user result against the standard of care laboratory test for HIV | Assessed at one time point only per patient (visit 1)approximately 1 hour
  The result obtained by the self-test user will be compared against a standard laboratory test for HIV
Comparison of self-test done in the laboratory against the standard of care laboratory blood test for HIV | Assessed at one time point only per patient (visit 1)approximately 1 hour
  The result obtained by a qualified lab technician using the participant's blood sample for the self-test will be compared against a standard laboratory blood test for HIV

CONTACTS AND LOCATIONS:
Overall Officials: Terrance J Thiel, Study Director — Atomo Diagnostics
Locations (1):
- Holdsworth House Medical Practice, Darlinghurst, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No